CLINICAL TRIAL: NCT06474559
Title: Comparison of Protector Laryngeal Mask With Endotracheal Tube: Evaluation of Respiratory Mechanical Parameters During Controlled Ventilation & Possibility of Pulmonary Aspiration
Brief Title: Comparison of Lma-Protector With Endotracheal Tube: Evaluation of Respiratory Mechanical Parameters During Controlled Ventilation & Possibility of Pulmonary Aspiration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Stella Antoniou, MD, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protector-1
Record Dates: First submitted 2024-06-05; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMA Protector (Experimental): LMA Protector will be inserted by a researcher after standard anesthesia induction. The view of the larynx will be assessed using fiberoptic grading scale. Mini bronchoalveolar lavage will be colected at the end of the procedure
  Interventions: Device: LMA Protector; Device: Endotracheal tube
- Endotracheal tube (Experimental): Patients will be intubated after standard anesthesia induction.The view of the larynx will be assessed ( Cormack Lehane system).Mini bronchoalveolar lavage will be colected at the end of the procedure
  Interventions: Device: LMA Protector; Device: Endotracheal tube

INTERVENTIONS:
Device: LMA Protector — LMA Protector will be inserted by a researcher after standard anesthesia induction. The view of the larynx will be assessed using fiberoptic grading scale.Mini bronchoalveolar lavage will be collected before the end of the procedure
Device: Endotracheal tube — tracheal intubation will be perform after standard anaesthetic induction. Cormack Lehane will be recorded. Mini bronchoalveolar lavage will be collected before the end of the procedure

SUMMARY:
The aim of this prospective, randomized, comparative, controlled clinical study is to compare laryngeal mask airway ProtectorTM with the endotracheal tube, regarding to the respiratory mechanical parameters during controlled mechanical ventilation and the prevalence of aspiration. Aspiration will be evaluated by detecting and quantifying pepsin (a marker of gastric aspiration) and α-amylase (a marker of salivary aspiration) in the bronchoalveolar lavage ( mini BAL) of patients ≥18 years old, ASA 1-2, undergoing selective low-risk surgery under general anesthesia in a lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years ASA1-2 who are to undergo planned urological surgery of low or intermediate severity, under general anesthesia in the lithotomy position.

Exclusion Criteria:

* patients < 18 years old.
* Patients who are going to undergo an emergency/urgent operation/ trauma patients.
* Maternal population.
* Patients who are not scheduled to receive general anesthesia, but some other type of anesthesia.
* Patients in whom LMA placement is contraindicated, such as patients at high risk for reflux and aspiration of gastric contents (eg, history of gastroesophageal reflux, hiatal hernia, pyloric stenosis, gastrointestinal obstruction, morbid obesity).
* Patients who meet at least one of the four RODS difficulty criteria.
* Contraindicated patients: administration of neuromuscular blockade, suppression of spontaneous respiration, and those with an indication for awake intubation or surgical airway.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Difference in PIP cmH20 (Peak inspiratory pressure ) between the two groups of patients. | Intraoperative
  Measured by Ventilator
Assessment of aspiration risk by quantitative measurements of pepsin (ng/ml) and α-amylase (IU/ml) in BAL of patients and differences in its incidence between the two groups. | through study completion, an average of 1 year
  Measured by ELISA method

SECONDARY OUTCOMES:
Differences in lung mechanics between the two patient groups | Intraoperative
  Pplat cmH20( plataeu pressure) Dynamic Compliance ml/cmH20 , MAP cmH20( Mean Airway pressure ), PEEP cmH20,( positive end-expiratory pressure VTins, VTexp ( t, Raw cmH20/ml/sec( resistance of airway), ΔP cmH20(Driving Pressure, inspired (VTinsp) and expired (VTexp) tidal volumes, VTins - VTexp.

CONTACTS AND LOCATIONS:
Locations (1):
- General Univerisity Hospital of Patras, Pátrai, Greece